CLINICAL TRIAL: NCT02698241
Title: Integrated Diagnostics Driven Diuretic and Chronic Medication Management for Heart Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INTERVENE-HF
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronization Therapy Defibrillator (CRT-D); heart failure; integrated diagnostics; chronic medication management
MeSH Terms: conditions — Heart Failure | interventions — Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic & Medication Management (Other): Enrolled subjects will be managed using integrated device diagnostics combined with a clinical medication plan.
  Interventions: Device: Diagnostic & Medication Management

INTERVENTIONS:
Device: Diagnostic & Medication Management — Single Arm Study. Subjects will be managed using integrated diagnostics.

SUMMARY:
The INTERVENE-HF study is a prospective, non-randomized, multi-center (US only), investigational, feasibility study. The purpose of this study is to characterize safety of managing heart failure patients with integrated device diagnostics that have an implanted commercially available Medtronic cardiac resynchronization therapy defibrillator (CRT-D).

DETAILED DESCRIPTION:
The study is expected to be conducted at up to 20 centers located in the United States. Up to 400 subjects will be enrolled to yield up to 200 eligible subjects that meet screening criteria. This study will be conducted in subjects with an implanted, commercially available, Medtronic, CRT-D device. Each enrolled subject will be followed every 2 months from time of enrollment to end of the study.The study will end after the last enrolled subject completes the 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject (or subject's legally authorized representative) is willing and able to provide written informed consent
* Subject has been implanted with a CRT device for at least 9 months and has had a wireless Medtronic CRT-D device for at least 34 days
* Subject has >1 year life expectancy
* Subject's CRT-D device has at least 18 months of device longevity left
* Subject has an eGFR> 25 ml/min/1.73 m2
* Subject is NYHA Class II or III
* Subject is NYHA Class II or III • Subject has elevated BNP values (BNP>400 or NTpro BNP>800) within the last 3 months OR Subject has had at least one OptiVol threshold crossing in the last 9 months OR Subject has had a HF event within the last 9 months

HF event is defined as meeting any one of the following two criteria:

1. Subject was admitted to the hospital for worsening HF OR
2. Subject has received Intravenous HF therapy (e.g. IV diuretics/vasodilators) or ultrafiltration at any settings including:

   * Emergency Department
   * Ambulance
   * Observation Unit
   * Urgent Care
   * HF/Cardiology Clinic
   * Patient's Home

     * Subjects who are currently prescribed and taking medications for the management of heart failure and are able to tolerate transient increases in diuretic dosage
     * Subject is willing and able to comply with the protocol, including screening, baseline and programming visit(s), remote care directions, follow-up visits, and exit visit
     * Subject can send device transmissions and daily biometric data with in-home patient devices

Exclusion Criteria

* Subject has systolic BP of < 90 mmHg at the time of enrollment
* Subject not responsive to diuretic therapy or is on chronic renal dialysis
* Subject unable to undergo one round of medication intervention (3 day up-titration of diuretic) without requiring safety check
* Subjects enrolled in a concurrent study that may confound the results of this study without documented pre-approval from a Medtronic study manager
* Subject weighs more than 500 pounds
* Subject is younger than 18 years of age
* Subject has hemodynamic monitoring device implanted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Warman, PhD, Study Director — Medtronic
Locations (8):
- United States (8):
  - Phoenix Cardiovascular Research Group, LLC, Phoenix, Arizona
  - Florida Heart Center, Ft. Pierce, Florida
  - Baptist Heart Specialists Research, Jacksonville, Florida
  - First Coast Cardiology, Jacksonville, Florida
  - South Miami Heart Specialists, Miami, Florida
  - Cardiology Partners, Wellington, Florida
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Lindner Research Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zile MR, Costanzo MRR, Ippolito EM, Zhang Y, Stapleton R, Sadhu A, Jimenez J, Hobbs J, Sharma V, Warman EN, Streeter L, Butler J. INTERVENE-HF: feasibility study of individualized, risk stratification-based, medication intervention in patients with heart failure with reduced ejection fraction. ESC Heart Fail. 2021 Apr;8(2):849-860. doi: 10.1002/ehf2.13231. Epub 2021 Feb 1. PMID 33527654

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A screening visit was required after a subject signed the informed consent form and before the baseline and programming visit. During the screening visit, subject's OptiVol Fluid Index and bloodwork were verified for the eligibility to continue the study. If subject failed the screening, he/she would exit the study.
Groups:
- Device Diagnostic & Diuretic and Chronic Medication Management: Enrolled subjects will be managed using integrated device diagnostics combined with a clinical medication plan. This is a single arm feasibility study.
Period: Overall Study
Arm/Group | Device Diagnostic & Diuretic and Chronic Medication Management
Started | 79 (Number of subjects enrolled the study)
Baseline & Programming (Subject characteristics collected and device diagnostic enabled at baseline and programming visit.) | 66 (Number of subjects that passed screening and completed baseline and programming visit)
Completed | 45 (Number of subjects completed the study (no early exit or death))
Not Completed | 34
Not completed — Inclusion/exclusion criteria not met | 4
Not completed — Screening not met | 7
Not completed — Withdrawal by Subject | 7
Not completed — Physician Decision | 2
Not completed — Subject underwent system modification | 2
Not completed — Lost to Follow-up | 3
Not completed — Subject on inodrip not safe to continue | 6
Not completed — geographic and licensing issue | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: After subjects passed the screening, they would attend the baseline & programming visit during which subjects' baseline characteristics was to be collected and OptiVol CareAlert should be turned on via device programming. Baseline analysis included subjects who passed the screening and completed the baseline & programming visit.
Arm/Group | Device Diagnostic & Diuretic and Chronic Medication Management
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 57
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 66
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.1 (6.4)
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 119.6 (17.7)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 70.6 (9.4)
NYHA Class [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification is commonly used to classify patients' heart failure according to the severity of their symptoms. It places patients in one of four categories based on how much they are limited during physical activity: Class I: No limitation of physical activity; Class II: Slight limitation of physical activity, comfortable at rest; Class III: Marked limitation of physical activity, comfortable at rest; Class IV: Unable to carry on any physical activity without discomfort. Higher classes mean worse conditions.
  Participants
    Class I | 0
    Class II | 27
    Class III | 39
    Class IV | 0
Having heart failure events in previous 6 months [Count of Participants; unit: Participants]
  Yes | 13
  No | 53

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of the Integrated Diagnostic Medication Intervention Strategy (i.e. Percentage of Implemented Interventions Being Effective)
Description: The Integrated Diagnostic Medication Intervention Strategy was physician-directed and nurse-implemented and it was based on a heart failure risk score diagnostic feature of a Medtronic CRT-D device implanted in the patients with heart failure. Effectiveness of this intervention strategy was measured as the percentage of implemented interventions being effective. Once initiated, an Integrated Diagnostic Medication Intervention would be effective if all the following criteria were met:
  1. The intrathoracic impedance of a subject recovered per defined criterion after completion of the Integrated Diagnostic Medication Intervention;
  2. The subject had no HF-related event (as adjudicated by the CEC) during or in the next 14 days after completion of the Integrated Diagnostic Medication Intervention;
  3. The subject had not experienced any adverse events that were related to the Integrated Diagnostic Medication Intervention per CEC adjudication and require medical care.
Time Frame: 12 months post enrollment
Population: All subjects who had received the Integrated Diagnostic Medication Intervention per protocol were in the scope of this endpoint analysis. The interest was the effectiveness of the implemented interventions.
Measure: Number; unit: percentage of effective interventions
Units Other Than Participants: Interventions Implemented
Arm/Group | Device Diagnostic & Diuretic and Chronic Medication Management
Number analyzed (Participants) | 66
Number analyzed (Interventions Implemented) | 26
percentage of effective interventions | 69.2

2. Primary Outcome: Safety of the Integrated Diagnostic and Medication Management (i.e. Percentage of Implemented Interventions Being Safe)
Description: The Integrated Diagnostic Medication Intervention Strategy was physician-directed and nurse-implemented and it was based on a heart failure risk score diagnostic feature of a Medtronic CRT-D device implanted in the patients with heart failure. Safety of this intervention strategy was measured as the percentage of implemented interventions being safe. Once initiated, the Integrated Diagnostic Medication Intervention Strategy would be regarded as being safe if all the following criteria were met:
  1. The Integrated Diagnostic Medication Intervention applied to an episode was not terminated due to safety issues;
  2. The Integrated Diagnostic Medication Intervention applied to an episode had not caused treatment-related adverse events (as adjudicated by the CEC).
Time Frame: 12 months post enrollment
Population: All subjects who had received the Integrated Diagnostic Medication Intervention per protocol were in the scope of this endpoint analysis. The interest was the safety of implemented interventions
Measure: Number; unit: percentage of safe interventions
Units Other Than Participants: Interventions Implemented
Arm/Group | Device Diagnostic & Diuretic and Chronic Medication Management
Number analyzed (Participants) | 66
Number analyzed (Interventions Implemented) | 26
percentage of safe interventions | 84.6

ADVERSE EVENTS:
Time Frame: In this study, adverse event data were collected from the time participants signed the informed consent to the time they died or completed the exit visit. The study planned to follow up subjects for 12 months.
Description: Only the following adverse events were monitored/assessed: all system-related adverse events (AEs), all cardiovascular-related AEs, all AEs that might be associated with the PRN intervention, and all serious adverse events (SAEs).
Arm/Group | Device Diagnostic & Diuretic and Chronic Medication Management
All-Cause Mortality (participants affected / at risk) | 2/79
Serious Adverse Events (participants affected / at risk) | 34/79
Other Adverse Events (participants affected / at risk) | 13/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Device Diagnostic & Diuretic and Chronic Medication Management (N=79)
Acute coronary syndrome (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Atrial flutter (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 10
Cardiac failure congestive (Cardiac disorders) | 6
Cardio-respiratory arrest (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Coronary artery stenosis (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Generalised oedema (General disorders) | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Pneumonia bacterial (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Device battery issue (Product Issues) | 1
Device lead damage (Product Issues) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Breast mass (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Air embolism (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Device Diagnostic & Diuretic and Chronic Medication Management (N=79)
Cardiac failure (Cardiac disorders) | 8
Hypotension (Vascular disorders) | 5

LIMITATIONS AND CAVEATS:
Enrollment was stopped after 79 patients were enrolled in the study and the preliminary safety interim data report was completed. The early stop was not due to any safety concerns. The sponsor deemed sufficient data had been collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT02698241/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT02698241/SAP_001.pdf